CLINICAL TRIAL: NCT01031537
Title: A Phase II, Open Label Trial of a Vaccine (FSME-IMMUN 0.5 mL) Against Tick-Borne Encephalitis (TBE) for NIAID Workers Manipulating Tick-Borne Encephalitis Virus (TBEV) in the Laboratory
Brief Title: Vaccine Study for Tick-Borne Encephalitis Virus (TBEV)
Acronym: TBEV
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Manufacturer discontinued support of the study
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 090246; 09-I-0246 (Other: National Institute of Allergy and Infectious Diseases)
Record Dates: First submitted 2009-12-11; First posted 2009-12-14 (Estimated); Results first posted 2018-07-05 (Actual); Last update posted 2018-07-05 (Actual); Status verified 2018-04

CONDITIONS: Tick-Borne Encephalitis; Encephalitis, Tick-Borne; Tick-Borne Disease; Glycoprotein E, Flavivirus; NSI Protein, Flavivirus
Keywords: FSME-Immun; TBEV; TBE Researcher; Plavivirus; Anti-TBEV Levels; Tic-Borne Encephalitis
MeSH Terms: conditions — Encephalitis, Tick-Borne; Tick-Borne Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FSME-IMMUN 0.5mL Baxter (Other): FSME-IMMUN 0.5mL Baxter is non-US licensed vaccine for tick-borne encephalitis virus. The FSME-IMMUN 0.5mL Baxter is available as 0.5mL in a pre-loaded vaccine syringe. All participants received active vaccine using a rapid immunization schedule, with vaccine administration on Days 0, 14, 161 and 245. Participants that tested seropositive for tick-borne encephalitis virus or subjects that developed positive viral neutralizer titers after the 3rd or 4th vaccine were given a booster of FSME-IMMUN 0.5mL Baxter vaccine at 3, 6 and 9 years after enrollment.
  Interventions: Biological: FSME-IMMUN 0.5ml Baxter

INTERVENTIONS:
Biological: FSME-IMMUN 0.5ml Baxter — Vaccine

SUMMARY:
This was an open label trial of a non-US licensed vaccine for tick-borne encephalitis. The vaccine was licensed by Baxter, and now following an acquisition by Pfizer Inc in Vienna, Austria since 2001, and has an extensive safety record in multiple European countries. Field effectiveness studies suggest > 99 percent protection against disease transmitted by the natural routes of either tick bite or ingestion of contaminated, unpasteurized milk. The vaccine is also considered to be effective against laboratory exposures and is used routinely for this purpose in European laboratories. The US Centers for Disease Control and Prevention and the National Institutes of Health acknowledge the effectiveness of the vaccine by allowing those who have received it to study tick-borne encephalitis virus (TBEV) in isolation facilities rated at BSL-3 rather than the more stringent BSL-4, with the exception of the Russian Spring-Summer Encephalitis strain. Subjects were recruited from personnel at 2 intramural campuses of the National Institute of Allergy and Infectious Diseases who may be exposed accidentally to any strain or serotype of viable TBEV. Approximately 160 individuals were eligible to participate. The rapid immunization schedule (injections on Days 0, 14, and 161) was used and subjects had labs drawn 21 days after the 2nd, 3rd and 4th vaccine injections to determine seroconversion. Subjects that seroconverted to TBEV were offered a booster dose of the vaccine 3 years from the date of receipt of the third dose of the vaccine. Subjects that were seropositive at entry into the study were offered a booster dose of the vaccine every 3 years from Day 0.

DETAILED DESCRIPTION:
Infection by tick-borne encephalitis virus (TBEV) is a significant health concern for humans in Europe and Asia. A vaccine is available in these regions and in Canada, but not in the United States. Research studies in Europe have shown the vaccine to be effective in preventing infection among the general population, where disease is transmitted either by the bite of an infected tick (most common) or by ingestion of contaminated unpasteurized milk or milk products. Persons who work with the virus in a research setting, however, have the potential of being exposed in unnatural ways, and may come into contact with concentrations of virus higher than those found naturally in ticks. The Food and Drug Administration is investigating the effectiveness of the existing vaccine. It is a killed vaccine, which means that it has been treated to ensure that it does not contain live agents (bacteria or virus). The manufacturer has tested the product for other possible contaminating agents and none have been detected. However, there is an unknown but small risk of exposure to undetected contaminating agents in the vaccine. This was an open label trial of a non-US licensed vaccine for tick-borne encephalitis. The vaccine has been licensed by Baxter, and now following an acquisition by Pfizer Inc in Vienna, Austria since 2001, and has an extensive safety record in multiple European countries. Field effectiveness studies suggest > 99 percent protection against disease transmitted by the natural routes of either tick bite or ingestion of contaminated, unpasteurized milk. The vaccine is also considered to be effective against laboratory exposures and is used routinely for this purpose in European laboratories. The US Centers for Disease Control and Prevention and the National Institutes of Health acknowledge the effectiveness of the vaccine by allowing those who have received it to study tick-borne encephalitis virus (TBEV) in isolation facilities rated at BSL-3 rather than the more stringent BSL-4, with the exception of the Russian Spring-Summer Encephalitis strain.

Subjects were recruited from personnel at 2 intramural campuses of the National Institute of Allergy and Infectious Diseases who may be exposed accidentally to any strain or serotype of viable TBEV. Approximately 160 individuals were eligible to participate.

Objectives: To test the safety and immune response to a vaccine against tick-borne encephalitis virus (TBEV). To add a level of protection to persons who may have occupational exposure to TBEV to reduce their chances of developing infection from that exposure.

Eligibility: Individuals 18 years of age or older who are in generally good health and have the potential for occupational exposure to TBEV at one of the two National Institute of Allergy and Infectious Diseases campuses.

Design: The full series of the vaccine included at least three doses by injection in the upper arm. The first and third dose of study vaccine were given in the muscle of the nondominant arm. The second dose was given in the dominant arm. Participation included at least 12 scheduled visits to the study center over approximately 3.5 years. An initial visit took place 7 to 21 days prior to the first injection. Blood samples were taken to test liver and kidney function, baseline antibody levels, and for possible pregnancy in female participants. Vaccine doses were given on days 0, 14, and 161. Participants were asked to complete a diary card on each day for one week following the vaccination to assess any reactions or side effects. At each visit after receipt of a vaccine, participants were asked about any side effects. Blood was drawn 14 days after the second injection and 21 days after the third injection in order to measure the level of antibodies and overall response to the vaccine. Subjects that developed a sufficiently high level of antibodies may (at the discretion of the laboratory chief) be allowed to work with strains of TBEV at Biosafety Level (BSL) 3 rather than BSL-4. Blood was drawn annually for 3 years to determine antibody level and response to the vaccine. Booster doses were provided if required.

ELIGIBILITY:
* INCLUSION CRITERIA:

All subjects must meet the following criteria at study entry:

* Be engaged in activities that place them at potential risk of occupational exposure to TBEV in its viable form at one of the participating intramural laboratories of NIAID
* Be 18 years of age or older at the time of the first immunization.
* Comprehend the study requirements.
* Provide written informed consent to participate in this study.
* Be in good health as determined by the Investigator, based upon medical history and a targeted physical examination.
* Have a stable health status as determined by the Investigator.
* Have access to a consistent means of telephone contact, which may be either in the home or at the workplace, land line or mobile, but NOT a pay phone or other multiple-user device (i.e., a common use phone serving multiple rooms or apartments).
* Express availability for the required study period, and ability to attend scheduled visits.

EXCLUSION CRITERIA:

The following criteria should be checked at the time of the study entry. If any apply, the subject will not be included in the study:

* The subject must not be participating in any other trial of an investigational drug or vaccine for 1 month prior to the first injection through until 21 days after the third injection. (Given the nature of the work these study subjects engage in, exemptions to this proscription may be granted on a case by case basis after discussion between the Investigator and the IRB.)
* The presence on the day of immunization of an oral temperature of >101.2 degrees F or acute symptoms other than mild severity.
* Active systemic infectious process as determined by review of systems and physical examination. The subject may be enrolled at a later date once the illness has resolved.
* Known immune suppression, such as that associated with human immunodeficiency virus infection, or other condition, to the extent that, in the opinion of the Investigator, the subject is likely to have a poor response to the vaccine. This information will be obtained by history only. Serologic screening for these diseases will not be performed.
* Presence of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if clinically stable, are deemed by the Investigator to render the potential subject unable/unlikely to report promptly any adverse reactions to the vaccine.
* Current diagnosis of leukemia, Hodgkin s disease, non-Hodgkin s lymphoma, or any other cancer, autoimmune disease such as lupus, which is in and of itself a cause of immunosuppression to the point that, in the opinion of the Investigator, the subject is likely to have a poor response to the vaccine.
* Currently receiving systemic immunosuppressive chemotherapy or immunotherapy (including glucocorticoids) resulting in immune suppression to the point that, in the opinion of the Investigator, the subject is likely to have a poor response to the vaccine.
* Any neurological condition in which (in the opinion of the Investigator) the integrity of the blood brain barrier may have been compromised.
* Licensed vaccines are not exclusionary but should be given at least 14 days before or after immunization (applies to each of the 3 scheduled TBEV injections) for inactivated vaccines and 30 days before or after immunization with any live vaccines. This is in order to avoid potential confusion of adverse reactions. (Given the nature of the work these study subjects engage in, exemptions to this proscription may be granted on a case-by-case basis after discussion between the Investigator and the IRB.).
* Previous anaphylactic reaction to any TBE vaccine.

Known or suspected anaphylactic reaction to any constituent of FSME IMMUN, to include formaldehyde, protamine sulfate, gentamicin and neomycin, or current egg allergy.

* Known pregnancy, or anticipating becoming pregnant in the first 8 months of the study or a positive urine beta-human chorionic gonadotropin (beta hCG) test result prior to immunization. If subjects become pregnant at some point in time after the 1st injection, no further injections will be given until after the pregnancy is completed, they are no longer nursing or have a negative beta-hCG result.
* Lactating or nursing.
* Women of child bearing potential (defined as pre-menopausal who have not undergone either hysterectomy or tubal ligation) who lack a history of reliable contraceptive practices. Reliable contraceptive practices (for the first 8 months of the study and within 21 days prior to or 42 days after booster immunizations) include:

  * Consistent abstinence from heterosexual activity
  * Consistent use of combined or progestogen oral contraceptives
  * Injectable progestogen
  * Implants of levonorgestrel
  * Estrogen or estrogen/progestogen vaginal ring
  * Percutaneous contraceptive patches
  * Intrauterine device (IUD) or intrauterine system (IUS)
  * Successful vasectomy of the sole male partner, or
  * Double barrier method (condom or occlusive cap plus spermicidal agent)
* A history of a prior infection with TBEV or previously receiving a TBE vaccine will not be considered as an exclusionary criterion for immunization through this protocol. However, these subjects antibody titer data will not be included in the statistical analysis.
* Any other conditions, which in the Investigator s judgment, might result in an increased risk to the subject, or would affect their participation in the study. Additionally the Investigator has the ability to exclude a subject if for any reason he/she feels the subject is not a good candidate for the study or will not be able to follow study procedures.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2009-09-25; Primary Completion 2016-12-23 (Actual); Study Completion 2016-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Schmitt, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Rocky Mountain Laboratory (RML), Hamilton, Montana

REFERENCES:
- [Background] Adner N, Leibl H, Enzersberger O, Kirgios M, Wahlberg T. Pharmacokinetics of human tick-borne encephalitis virus antibody levels after injection with human tick-borne encephalitis immunoglobulin, solvent/detergent treated, FSME-BULIN S/D in healthy volunteers. Scand J Infect Dis. 2001;33(11):843-7. doi: 10.1080/00365540110027358. PMID 11760166
- [Background] Baumhackl U, Franta C, Retzl J, Salomonowitz E, Eder G. A controlled trial of tick-borne encephalitis vaccination in patients with multiple sclerosis. Vaccine. 2003 Apr 1;21 Suppl 1:S56-61. doi: 10.1016/s0264-410x(02)00815-0. PMID 12628815
- [Background] Charrel RN, Attoui H, Butenko AM, Clegg JC, Deubel V, Frolova TV, Gould EA, Gritsun TS, Heinz FX, Labuda M, Lashkevich VA, Loktev V, Lundkvist A, Lvov DV, Mandl CW, Niedrig M, Papa A, Petrov VS, Plyusnin A, Randolph S, Suss J, Zlobin VI, de Lamballerie X. Tick-borne virus diseases of human interest in Europe. Clin Microbiol Infect. 2004 Dec;10(12):1040-55. doi: 10.1111/j.1469-0691.2004.01022.x. PMID 15606630

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects withdrew after the screening visit and elected not re-enroll. 1 subject was a study screen failure.
Groups:
- FSME-IMMUN 0.5mL Baxter: FSME-IMMUN 0.5mL Baxter is non-US licensed vaccine for tick-borne encephalitis. The FSME-IMMUN 0.5mL Baxter is available as 0.5mL in a pre-loaded vaccine syringe. All participants will receive active vaccine using a rapid immunization schedule, with vaccine administration on Days 0, 14, 161 and 245. Participants that test seropositive for tick-borne encephalitis or subjects that develop positive viral neutralizer titers after the 3rd or 4th vaccine will be given a booster of FSME-IMMUN 0.5mL Baxter vaccine at 3, 6 and 9 years after enrollment.
  FSME-IMMUN 0.5ml Baxter: Vaccine
Period: Overall Study
Arm/Group | FSME-IMMUN 0.5mL Baxter
Started | 66
Completed | 34
Not Completed | 32
Not completed — medical reasons not related to study | 3
Not completed — Lack of Efficacy | 1
Not completed — retired from NIH, met exclusion criteria | 1
Not completed — moved, met exclusion criteria | 10
Not completed — Withdrawal by Subject | 5
Not completed — PI removal, no longer met eligibility | 12

BASELINE CHARACTERISTICS:
Groups:
- FSME-IMMUN 0.5mL Baxter: FSME-IMMUN 0.5mL Baxter is non-US licensed vaccine for tick-borne encephalitis. The FSME-IMMUN 0.5mL Baxter is available as 0.5mL in a pre-loaded vaccine syringe. All participants received active vaccine using a rapid immunization schedule, with vaccine administration on Days 0, 14, 161 and 245. Participants that tested seropositive for tick-borne encephalitis or subjects that developed positive viral neutralizer titers after the 3rd or 4th vaccine were given a booster of FSME-IMMUN 0.5mL Baxter vaccine at 3, 6 and 9 years after enrollment.
  FSME-IMMUN 0.5ml Baxter: Vaccine
Arm/Group | FSME-IMMUN 0.5mL Baxter
Number analyzed (Participants) | 66
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 66
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 4
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 66
Tick-Borne Encephalitis Virus Antibody Neutralization Titer [Count of Participants; unit: Participants] — Tick-Borne Encephalitis Virus Neutralization antibody level is a laboratory test collected via peripheral venipuncture.
  Titer levels > 1:10 reflect the presence of protective antibodies to Tick-Borne Encephalitis Virus.
  Presence of protective antibody titers at baseline indicate either prior successful immunization or previous infection from Tick-Borne Encephalitis Virus.
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: TBEV Viral Neutralization Titer >1:10
Description: Tick borne encephalitis antibody viral neutralization titer levels (>1:10)
Time Frame: Baseline
Population: Baseline TBEV protective antibody levels (>1:10) reflective of either prior successful immunization or infection at baseline
Measure: Count of Participants; unit: Participants
Arm/Group | FSME-IMMUN 0.5mL Baxter
Number analyzed (Participants) | 66
Participants | 6

2. Primary Outcome: TBEV Viral Neutralization Titer >1:10
Description: The number of participants that develop anti-tick borne encephalitis antibody viral neutralization titer levels (>1:10) following receipt of 3 doses of intramuscular FSME-IMMUN (vaccine series)
Time Frame: 6 months
Population: Six participants had protective antibody levels (>1:10) reflective of either prior successful immunization or infection at baseline and were not evaluated at the 6 month time point. One participant withdrew from the study prior to the 6 month evaluation time point.
Measure: Count of Participants; unit: Participants
Arm/Group | FSME-IMMUN 0.5mL Baxter
Number analyzed (Participants) | 59
Participants | 58

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from baseline (day 0), and on days 7, 14, 21, 35, 161, 168, 182, 245, 252, and 266, 3 years, and up to 6 years after vaccination. Note study was prematurely closed on July 5, 2016 as the manufacturer elected to stop providing the vaccine support for this study.
Arm/Group | FSME-IMMUN 0.5mL Baxter
All-Cause Mortality (participants affected / at risk) | 0/66
Serious Adverse Events (participants affected / at risk) | 10/66
Other Adverse Events (participants affected / at risk) | 64/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSME-IMMUN 0.5mL Baxter (N=66)
Pulmonary granuloma (Respiratory, thoracic and mediastinal disorders) | 1
Urinary tract infection, relapsing fever (Infections and infestations) | 2
Bladder laceration (Injury, poisoning and procedural complications) | 1
Ovarian cyst (Reproductive system and breast disorders) | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Stage IV lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Uterine fibroid (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FSME-IMMUN 0.5mL Baxter (N=66)
Pain at the injection site (Musculoskeletal and connective tissue disorders) | 64
Headache (Nervous system disorders) | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 18
Fatigue (General disorders) | 19
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Swelling (Skin and subcutaneous tissue disorders) | 1
Itching (Skin and subcutaneous tissue disorders) | 1
Bruising (Skin and subcutaneous tissue disorders) | 1
Malaise (General disorders) | 1
Chills (General disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes